CLINICAL TRIAL: NCT04611269
Title: Clinical Characteristics and Outcomes of Patients With COVID-19 on Mechanical Ventilation in Argentina: a Prospective, Multicenter Cohort Study
Brief Title: Clinical Characteristics and Outcomes of Patients With COVID-19 on Mechanical Ventilation in Argentina
Acronym: SATICOVID19
Status: Completed | Type: Observational
Sponsor: Argentinian Intensive Care Society (Other)
Responsible Party: Principal Investigator, Elisa Estenssoro, MD, Argentinian Intensive Care Society
Other Study IDs: SATI
Record Dates: First submitted 2020-10-29; First posted 2020-11-02 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Respiratory Failure; Covid-19; Mechanical Ventilation
MeSH Terms: conditions — Respiratory Insufficiency; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult, patients with COVID-19 admitted to the ICU requiring mechanical ventilation: This is a prospective cohort study including patients >18 years RT-PCR positive for SARS Cov-2 admitted to the ICU that require mechanical ventilation. Epidemiological data, comorbidities, previous signs of symptoms of COVID-19. On admission, severity of disease scores, laboratory management data, blood gases and acid-base chemistry,respiratory and mechanical ventilation management,and complications (Development of ARDS, septic shock, acute kidney injury, thromboembolic events, infections and septic shock, will be recorded. If patients die, causes of death will be recorded.Treatments administered by attending physicians will be registered.
  Dates of hospital and ICU admission, of death and/or discharge will be recorded.
  No intervention will be administered. Follow-up will continue until death or ICU/hospital discharge

SUMMARY:
The main objective of the present study is to determine ICU and in-hospital mortality associated with COVID-19 infection and its independent predictors, in patients admitted to adult ICUs in Argentina with a requirement for mechanical ventilation.

Secondary objectives include: determining epidemiological and clinical data in patients with COVID-19 disease; the associated morbidity, the support and therapeutic measures implemented, and the evolution of these patients upon discharge from the ICU.

Likewise, characteristics of each ICU will be recorded, and a survey will be carried out on the management of the COVID-19 pandemic, which will require information on the additional availability of critical resources for the care of patients admitted to the ICU. Likewise, characteristics of the ICU and hospitals will be registered.

DETAILED DESCRIPTION:
In December 2019, China reported cases of acute respiratory disease caused by a new beta-coronavirus (SARS-CoV-2), called COVID-19 by the WHO. In January 2020 this entity issues an alert about the emergence of this new disease throughout the world, and in March it declares it a pandemic. Severe cases represent around 14-20% of those reported, and admission to the ICU is highly variable according to the different publications and severity of disease, ranging between 29% and 89%. The mortality reported in these publications ranges between 1.4 and 42%; with the development of acute respiratory distress syndrome (ARDS) being one of the most severe complications, associated with worst outcomes. However, the time of appearance of symptoms of severe acute respiratory failure has shown significant variability between these studies, with a median appearance of 2, 5 and 14 days from the onset of symptoms of the disease.

As of March 21, 2020, cases in Latin America were increasing, finding countries such as Brazil, Chile, Ecuador, Peru and Argentina among the countries with the highest number of confirmed cases, being classified as countries with local transmission. Since there is no information about on the behavior of this new disease in our country, the Argentine Society of Intensive Care (SATI) launched an epidemiological study to know the characteristics, risk factors and evolution of the most severely compromised patients with COVID-19, those admitted to the ICU requiring mechanical ventilation (MV).

Therefore, the main objective of the present study is to determine the ICU and in-hospital mortality associated with COVID-19 infection and its independent predictors, in patients admitted to adult ICUs in Argentina on MV.

Secondary objectives include: determining epidemiological and clinical data and mechanical ventilation management in patients with COVID-19 , support and therapeutic measures implemented by their assistant physicians, and the evolution and complications developed by these patients during their ICU stay. The different causes of death will also be recorded.

Likewise, characteristics of each ICU will be recorded, and a survey will be carried out on the management of the COVID-19 pandemic, which will require information on the additional availability of critical resources for the care of patients admitted to the ICU. The opinion about the management of the pandemic by the different governmental strata will be required, in order to detect possible points of improvement in the external management of the pandemic.

ELIGIBILITY:
Inclusion Criteria:

- Consecutive adult patients admitted to participating ICUs who require mechanical ventilation and present confirmed COVID-19 .

Exclusion Criteria:

* Patients with severe respiratory infections / pneumonia due to another proven etiology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Confirmed case:
  Any suspected or probable case that presents positive results by rtPCR for SARS CoV-2.
Sampling Method: Non-Probability Sample
Enrollment: 950 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
ICU Mortality | From inclusion up to 90 days.
  Refers to patients dying during their stay at the ICU, whatever the cause

SECONDARY OUTCOMES:
Hospital mortality | From date of inclusion to date of death from any cause, assessed up to 90 days
  Refers to patients dying in the hospital, whatever the cause, after ICU discharge

OTHER OUTCOMES:
Independent predictors of mortality | Through study completion, up to 90 days
  Variables independently associated with mortality, according to multivariable analysis
Length of invasive mechanical ventilation | From date of intubation day to date of definitive weaning (more than 48 hours without the need of mechanical ventilation)
  Days on invasive mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Estenssoro, MD, Study Chair — Hospital Interzonal de Agudos San Martin de La Plata
Locations (5):
- Argentina (5):
  - Hospital Interzonal General de Agudos Gral. San Martín, La Plata, Buenos Aires
  - Sanatorio Las Lomas, San Isidro, Buenos Aires
  - Hospital General de Agudos Juan A. Fernández, Buenos Aires, Buenos Aires F.D.
  - Sanatorio Anchorena Recoleta, Buenos Aires, Buenos Aires F.D.
  - Sanatorio Otamendi, Buenos Aires, Buenos Aires F.D.

IPD SHARING:
Plan to Share IPD: Yes
Data on duration of mechanical ventilation, ICU and Hospital stay will be shared
Supporting Information: CSR
Time Frame: Data from patients included from April 30 to August 1, 2020, will be shared between October 1 and December 2020
Access Criteria: Data needed to perform mathematical models about duration of mechanical ventilation and ICU and hospital stay

REFERENCES:
- [Result] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Result] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Result] Wu C, Chen X, Cai Y, Xia J, Zhou X, Xu S, Huang H, Zhang L, Zhou X, Du C, Zhang Y, Song J, Wang S, Chao Y, Yang Z, Xu J, Zhou X, Chen D, Xiong W, Xu L, Zhou F, Jiang J, Bai C, Zheng J, Song Y. Risk Factors Associated With Acute Respiratory Distress Syndrome and Death in Patients With Coronavirus Disease 2019 Pneumonia in Wuhan, China. JAMA Intern Med. 2020 Jul 1;180(7):934-943. doi: 10.1001/jamainternmed.2020.0994. PMID 32167524
- [Result] Docherty AB, Harrison EM, Green CA, Hardwick HE, Pius R, Norman L, Holden KA, Read JM, Dondelinger F, Carson G, Merson L, Lee J, Plotkin D, Sigfrid L, Halpin S, Jackson C, Gamble C, Horby PW, Nguyen-Van-Tam JS, Ho A, Russell CD, Dunning J, Openshaw PJ, Baillie JK, Semple MG; ISARIC4C investigators. Features of 20 133 UK patients in hospital with covid-19 using the ISARIC WHO Clinical Characterisation Protocol: prospective observational cohort study. BMJ. 2020 May 22;369:m1985. doi: 10.1136/bmj.m1985. PMID 32444460
- [Result] Ferrando C, Suarez-Sipmann F, Mellado-Artigas R, Hernandez M, Gea A, Arruti E, Aldecoa C, Martinez-Palli G, Martinez-Gonzalez MA, Slutsky AS, Villar J; COVID-19 Spanish ICU Network. Clinical features, ventilatory management, and outcome of ARDS caused by COVID-19 are similar to other causes of ARDS. Intensive Care Med. 2020 Dec;46(12):2200-2211. doi: 10.1007/s00134-020-06192-2. Epub 2020 Jul 29. PMID 32728965
- [Result] Wunsch H. Mechanical Ventilation in COVID-19: Interpreting the Current Epidemiology. Am J Respir Crit Care Med. 2020 Jul 1;202(1):1-4. doi: 10.1164/rccm.202004-1385ED. No abstract available. PMID 32402207
- [Result] Bouadma L, Lescure FX, Lucet JC, Yazdanpanah Y, Timsit JF. Severe SARS-CoV-2 infections: practical considerations and management strategy for intensivists. Intensive Care Med. 2020 Apr;46(4):579-582. doi: 10.1007/s00134-020-05967-x. Epub 2020 Feb 26. No abstract available. PMID 32103284
- [Derived] Estenssoro E, Loudet CI, Rios FG, Kanoore Edul VS, Plotnikow G, Andrian M, Romero I, Piezny D, Bezzi M, Mandich V, Groer C, Torres S, Orlandi C, Rubatto Birri PN, Valenti MF, Cunto E, Saenz MG, Tiribelli N, Aphalo V, Reina R, Dubin A; SATI-COVID-19 Study Group. Clinical characteristics and outcomes of invasively ventilated patients with COVID-19 in Argentina (SATICOVID): a prospective, multicentre cohort study. Lancet Respir Med. 2021 Sep;9(9):989-998. doi: 10.1016/S2213-2600(21)00229-0. Epub 2021 Jul 2. PMID 34224674